CLINICAL TRIAL: NCT03500640
Title: Reducing Cardiometabolic Risk and Promoting Functional Health in Community-based Elders With Obesity and Pre-diabetes: Evaluating Sustainable DPP Follow-up Strategies
Brief Title: Reducing Cardiometabolic Risk and Promoting Functional Health in Older Adults With Obesity and Prediabetes
Acronym: Sustain-DPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Venditti, Associate Professor of Psychiatry and Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO17060604; R01DK114115 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-04-18 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Obesity; PreDiabetes; Aging
Keywords: Intervention; Prevention; Weight Management; Physical Activity; Physical Function
MeSH Terms: conditions — Obesity; Prediabetic State; Motor Activity

STUDY DESIGN:
Intervention Model Description: An initial 16-session Diabetes Prevention Program (DPP), called Group Lifestyle Balance (GLB) and aligned with current Medicare guidelines, will be administered to all enrolled participants primarily through group telephone contact, videos, and workbooks. Subsequently one-half of those enrolled will be randomly assigned to either (1) 30-minute DPP behavior intervention group telephone contact, or (2) 15-minute support group telephone contact for a total of 18 additional follow up months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPP Plus 30-minute calls (Active Comparator): Following the 6-month, 16-session, DPP core program, 30-minute group telephone calls will be implemented. Structured behavioral DPP maintenance sessions with a healthy aging focus occur once-per-month from months 7 to 12, and every-two-months from months 13 to 24.
  Interventions: Behavioral: DPP Intensive: 30-minute calls
- DPP Minimal 15-minute calls (Placebo Comparator): Following the 6-month, 16-session, DPP core program, 15-minute group telephone calls will be implemented. Social-support sessions occur once-per-month from months 7 to 12, and every-two-months from months 13 to 24.
  Interventions: Behavioral: DPP Support: 15-minute calls

INTERVENTIONS:
Behavioral: DPP Intensive: 30-minute calls — Ongoing DPP intervention and behavioral progress review to prevent relapse and improve cardiometabolic and functional health targets as keys to healthy aging.
  Other Names: Behavior Change/Relapse Prevention/Healthy Aging
  Arms: DPP Plus 30-minute calls
Behavioral: DPP Support: 15-minute calls — No further behavioral intervention materials provided; phone-contacts for mutual social support and accountability
  Other Names: Social Support
  Arms: DPP Minimal 15-minute calls

SUMMARY:
Obesity and pre-diabetes threatens the overall health and functional independence of older adults but lifestyle weight management for diabetes prevention, soon to be reimbursed by Medicare, can reduce this burden. The current 24-month study will enroll adults, ages 60 and older, through senior community centers and research registries. The investigators will study how two long term weight loss maintenance programs, both using group telephone sessions to support health behavior change, impact meaningful health outcomes. If successful, this project will provide a sustainable intervention model for healthy aging services that can benefit older adults and society.

DETAILED DESCRIPTION:
The confluence of obesity and pre-diabetes in older adults increases the risk of diabetes, and accelerates functional decline, chronic disease, disability, and death. More research is needed to refine and extend preventive interventions to reduce burden for vulnerable individuals and society. For over a decade efficacious 6- and 12-month Diabetes Prevention Program (DPP) lifestyle interventions have been translated successfully and shown positive impact. However, efforts to develop and evaluate scalable programs conforming to current guidelines for longer term DPP interventions (up to 24 months), which are consistent with a chronic care model, and help a greater proportion of enrollees sustain the recommended weight loss target of ≥ 5% are lacking. The scientific premise is that evaluation of translational DPP interventions, which has centered largely on strategies for weight loss induction, must be extended to include scalable longer-term interventions that show meaningful weight, cardiometabolic and functional health benefits for vulnerable older adults in community-based settings. A previous DPP-based study from this group of investigators documented the utility of telephone follow-up after 12-weeks of DPP weight loss induction and demonstrated that 63% of the 65-80-year-old volunteer sample with obesity and other risk factors were able to sustain ≥ 5% weight loss at 12-months. Despite good evidence that longer duration lifestyle interventions yield better outcomes (reflected in the latest Medicare ruling) there are no translational studies of 24-month long DPP-based interventions for older adults exclusively. The investigators will recruit participants from a broad array of community settings and examine how best to sustain the impact of a healthy lifestyle-healthy aging focused DPP with scalable treatment components over a 24-month period. The Sustain-DPP study will recruit and enroll adults 60 years of age and older, with overweight/obesity (BMI >= 27) and pre-diabetes (either HbA1c of 5.7 to 6.4% inclusive or fasting glucose >=100 but less than 126 mg/dL) (N = 360) from a network of community centers that offer healthy aging services and from community research registries. The intervention program sequence has been designed to align with current Medicare guidelines. First, from 0-6 months, experienced lifestyle coaches will administer a combination of in-person, video and telephone coaching sessions for all participants, at least 25% from ethnic/racial minority groups. Next, individual participants will be randomized (N = 180 per arm; stratified by weight loss of < or ≥ 5% and other demographic factors) to one of two 18-month follow-up conditions delivered as once-a-month telephone sessions only from 6-24 months. The investigators will compare the effects of (1) 30-minute behavioral intervention sessions, which include a Medicare-DPP and healthy lifestyle for healthy aging focus, and (2) 15-minute social support sessions, on measures of weight (the primary outcome) at 12-, 18-, and 24-months. In addition, data will be collected on cardiometabolic, physical activity, physical function, psychosocial, behavioral and other age-sensitive quality of life measures at 12- and 18- and 24-months. Finally, Medicare claims data will be examined for a proportion of the sample regarding medication use, outpatient, inpatient, and emergency visits and enrollment/participation in elder-focused activity programs. This work, if successful, will have immediate potential for DPP-sustainable lifestyle interventions that benefit vulnerable aging individuals and society.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Ages 60 and older
* Body mass index (BMI) >= 27 kg/m2
* Prediabetes defined as Hemoglobin (HbA1c) >= 5.7 % and <= 6.4 % or fasting glucose of >= 100 mg/dL and less than 126 mg/dL (at either screening or baseline visit)
* Access to a telephone (for group calls) and to video-player or computer with Internet (to watch session videos and activity videos)
* Able to travel to one of the community clinics in Southwestern Pennsylvania to participate in the first four in-person intervention sessions and five health assessments at 0, 6, 12, 18, and 24 months
* Has health care provider permission to participate

Exclusion Criteria:

* Currently diagnosed with diabetes (defined as HbA1c of >= 6.5% at either screening or baseline visit)
* Currently taking glucose lowering medications or weight loss medications
* Weight loss of 9 pounds or more in the last six months
* History of bariatric surgery within the last 2 years
* Permanently confined to wheelchair
* Significant cognitive or psychiatric disability that would preclude participation in normal community-based educational activities

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Venditti, PhD, Principal Investigator — Univ. Pittsburgh School of Medicine-Dept. Psychiatry
Locations (1):
- Univ. Pittsburgh School of Medicine-Dept. Psychiatry, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will follow the guidance of NIDDK on data preparation and sharing policies and insure there is permission to disclose de-identified individual participant-level data collected prior to releasing it to other researchers. In addition, requesting researchers must meet all NIDDK access requirements. Study investigators will maintain strict compliance with Human Research Protections/IRB requirements and use appropriate safeguards before sharing any IPD with other researchers. Within 3 years following final data collection, the investigators will prepare and share the final, completely de-identified dataset (IPD) with NIDDK to be made available to other researchers. However, the investigators will not share other statistical code or data dictionaries.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years from the final data collection of the last participant
Access Criteria: Investigators will share data through the NIDDK central repository (website shown below)
URL: http://repository.niddk.nih.gov/home/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After working with key stakeholders in the community, the study start date was March 27, 2018, and recruitment continued through February 2021. Recruitment was conducted in six waves, focusing on public and private senior centers and recreation facilities, senior residences, church ministries, medical practices, and senior/retiree database registries. Methods included in-person presentations, newspaper and digital media blasts, and direct-mail postcards.
Pre-assignment Details: Of 314 participants enrolled, all were offered a base 16-session DPP intervention (0-6 months) through group teleconference contact, videos, and workbooks. Of these, 258 participants were randomized to the two-group teleconference follow-up contact arms. Although the "Period 1" 0-6-month outcomes data will be reported in the final outcomes' manuscript, these pre-randomization data are not intended to be part of the primary or secondary analyses.
Groups:
- DPP Core Program: In Period 1, from 0-6 months, the DPP Core Program was implemented for ALL participants (pre-randomization). The DPP Core Program consisted of the base 16-session DPP intervention delivered through group teleconference contact, self-directed videos, and workbooks
- DPP Plus: 30 Minute Calls: In Periods 2, 3, and 4, DPP Plus: 30-minute calls were implemented (post-randomization). These consisted of structured behavioral DPP maintenance sessions with a healthy aging focus. Sessions occurred once-per-month (7-12 months) then every two months (13-16 months and 18-24 months). The ongoing DPP intervention sessions were designed to be behaviorally intensive and provided behavioral goals review and new learning materials at each contact.
- DPP Minimal: 15-Minute Calls: In Periods 2, 3, and 4, DPP Minimal: 15-Minute Calls were implemented (post-randomization). These were coach-introduced and facilitated but consisted primarily of unstructured peer discussion. Sessions occurred once-per-month (7-12 months) then every two months (13-16 months and 17-24 months) parallel to the DPP-30-minute arm. These intervention sessions were designed to promote peer support and accountability and no new learning materials were provided.
Period: DPP Core Program (0-6 Months)
Arm/Group | DPP Core Program | DPP Plus: 30 Minute Calls | DPP Minimal: 15-Minute Calls
Started | 314 | 0 | 0
Completed | 258 | 0 | 0
Not Completed | 56 | 0 | 0
Not completed — Lost to Follow-up | 26 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 0 | 0
Not completed — No Exercise Clearance | 3 | 0 | 0
Not completed — Spouses (Per Protocol) Excluded | 6 | 0 | 0
Period: Follow-Up Contacts (7-12 Months)
Arm/Group | DPP Core Program | DPP Plus: 30 Minute Calls | DPP Minimal: 15-Minute Calls
Started (The DPP Core Program intervention ended at 6 months, per protocol.) | 0 | 129 | 129
Completed (The DPP Core Program intervention ended at 6 months, per protocol.) | 0 | 95 | 84
Not Completed | 0 | 34 | 45
Not completed — Lost to Follow-up | 0 | 33 | 41
Not completed — Withdrawal by Subject | 0 | 1 | 4
Period: Follow-up Contacts (13-18 Months)
Arm/Group | DPP Core Program | DPP Plus: 30 Minute Calls | DPP Minimal: 15-Minute Calls
Started (The DPP Core Program intervention ended at 6 months, per protocol.) | 0 | 95 | 84
Completed | 0 | 93 | 74
Not Completed | 0 | 2 | 10
Not completed — Lost to Follow-up | 0 | 1 | 9
Not completed — Withdrawal by Subject | 0 | 1 | 1
Period: Follow-Up Contacts (19-24 Months)
Arm/Group | DPP Core Program | DPP Plus: 30 Minute Calls | DPP Minimal: 15-Minute Calls
Started (A final Wave 6 cohort (n = 25 assigned to DPP Plus and n = 13 assigned to DPP Minimal) were enrolled in PIVOT with a priori knowledge that only 18 months of study follow-up was possible.) | 0 | 68 | 61
Completed | 0 | 65 | 60
Not Completed | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: DPP Plus: 30-minute Calls: Behavioral: DPP Intensive 30-minute calls include ongoing DPP intervention. Structured, workbook-based maintenance sessions with a healthy aging focus occur once-per-month from months 7 to 12, and every-two-months from months 13 to 24.
- Placebo Comparator: DPP Minimal: 15-minute Calls: Behavioral: DPP Support 15-minute calls include no further behavioral intervention or self-monitoring materials; phone contacts are unstructured and intended to enhance peer support and accountability.
- Total: Total of all reporting groups
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [64 to 72] | 67 [64 to 71] | 68 [64 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 42 | 43 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  non-Hispanic Black or Black/Mixed Race | 21 | 19 | 40
  non-Hispanic White | 108 | 109 | 217
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Body mass index (BMI) is a measure of bodyfat based on height and weight. BMI is calculated as average weight divided by average height squared (kg/m2). In the clinic, height is measured in street clothes, without shoes, using a Shorr wall-mounted stadiometer. Weight is taken twice and measured to the nearest 0.1 kg using a SECA 880 digital scale.
  kg/m2 | 35.5 (5.6) | 35.4 (6.1) | 35.4 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bodyweight
Description: Percent bodyweight change (clinic measured) of participant
Time Frame: 12-month change from baseline bodyweight
Population: 129 participants were randomized to the Active Comparator and 129 were randomized to the Placebo Comparator at 6-months. Although self-reported weights were obtained, the analytic sample here is ONLY for those with objective clinic measured bodyweight data. This was available for 95 (74%) of Active Comparator and 84 (65%) of the Placebo Comparator arms at 12-months.
Measure: Mean (95% Confidence Interval); unit: percentage of bodyweight change
Groups:
- Active Comparator: DPP Plus 30-minute Calls: DPP Behavioral Intensive 30-minute calls include ongoing DPP intervention. Structured, workbook-based maintenance sessions with a healthy aging focus occur once-per-month from months 7 to 12, and every-two-months from months 13 to 24.
- Placebo Comparator: DPP Minimal 15-minute Calls: DPP Support 15-minute calls include no further behavioral intervention or self-monitoring material; phone contacts are unstructured and designed to promote peer support and accountability.
Arm/Group | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
Number analyzed (Participants) | 95 | 84
percentage of bodyweight change | -7.4 [-8.9 to -5.9] | -6.1 [-7.4 to -4.7]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus 30-minute Calls vs Placebo Comparator: DPP Minimal 15-minute Calls; Test type: Superiority; p = 0.196, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05

2. Primary Outcome: Change in Bodyweight
Description: Percent bodyweight change (clinic measured) of participant
Time Frame: 18-month change from baseline bodyweight
Population: 129 participants were randomized to the Active Comparator and 129 were randomized to the Placebo Comparator at 6-months. Although self-reported weights were obtained, the analytic sample here is ONLY for those with objective clinic measured bodyweight data. Of these, clinic measured bodyweight data was available for 93 (72%) of Active Comparator and 74 (57%) of the Placebo Comparator arms at 18-months.
Measure: Mean (95% Confidence Interval); unit: percent bodyweight change
Arm/Group | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
Number analyzed (Participants) | 93 | 74
percent bodyweight change | -6.4 [-8.0 to -4.7] | -6.1 [-7.7 to -4.4]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus 30-minute Calls vs Placebo Comparator: DPP Minimal 15-minute Calls; Test type: Superiority; p = 0.800, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05

3. Primary Outcome: Change in Bodyweight
Description: Percent bodyweight change (clinic measured) of participant.
Time Frame: 24-month change from baseline bodyweight
Population: 129 participants were randomized to the Active Comparator and 129 were randomized to the Placebo Comparator at 6-months. Although self-reported weights were obtained, the analytic sample here is ONLY for those with objective clinic measured bodyweight data. Of these, clinic measured bodyweight data was available for 65 (50%) of the Active Comparator and 60 of Placebo Comparator (46.5%) arms at 24-months.
Measure: Mean (95% Confidence Interval); unit: percent bodyweight change
Arm/Group | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
Number analyzed (Participants) | 65 | 60
percent bodyweight change | -4.6 [-6.2 to -3.1] | -5.1 [-6.8 to -3.4]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus 30-minute Calls vs Placebo Comparator: DPP Minimal 15-minute Calls; Test type: Superiority; p = 0.677, t-test, 2 sided

4. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference measured in centimeters with a Gulick spring-loaded tape measure.
Time Frame: 12-month.change from baseline waist circumference
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 95 | 84
centimeters | -6.0 [-7.6 to -4.5] | -4.6 [-7.3 to -1.9]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.349, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05

5. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference measured in centimeters with a Gulick spring-loaded tape measure.
Time Frame: 24-month change from baseline waist circumference
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 60
centimeters | -2.2 [-3.9 to -0.5] | -2.5 [-6.1 to 1.2]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.891, t-test, 2 sided

6. Secondary Outcome: Change in Fasting Glucose
Description: Fasting glucose (mg/dL) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens were analyzed at a central research laboratory.
Time Frame: 12-month change from baseline fasting glucose
Population: The analytic sample here represents only those for whom a valid laboratory test was obtained. No imputation methods were used.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 66 | 55
mg/dL | -5.3 [-7.9 to -2.6] | -2.3 [-5.3 to 0.6]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.140, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05

7. Secondary Outcome: Change in Fasting Glucose
Description: Fasting glucose (mg/dL) blood samples will be taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens are analyzed at a central research laboratory.
Time Frame: 24-month change from baseline fasting glucose
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 56 | 43
mg/dL | -4.2 [-7.2 to -1.1] | -4.9 [-8.2 to -1.7]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.732, t-test, 2 sided

8. Secondary Outcome: Change in Fasting Insulin
Description: Fasting insulin blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens were analyzed at a central research laboratory. All collected data values obtained will be converted for uniformity to pmol/L.
Time Frame: 12-month change from baseline fasting insulin
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
Number analyzed (Participants) | 71 | 53
pmol/L | -21.3 [-31.7 to -10.9] | -17.6 [-29.4 to -5.7]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus 30-minute Calls vs Placebo Comparator: DPP Minimal 15-minute Calls; Test type: Superiority; p = 0.637, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05

9. Secondary Outcome: Change in Fasting Insulin
Description: as for outcome 8
Time Frame: 24-month change from baseline fasting insulin
Population: The analytic sample here represents only those for whom a valid laboratory test was performed.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
Number analyzed (Participants) | 53 | 44
pmol/L | -16.8 [-29.4 to -4.1] | -8.5 [-25.3 to 8.3]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus 30-minute Calls vs Placebo Comparator: DPP Minimal 15-minute Calls; Test type: Superiority; p = 0.521, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05

10. Secondary Outcome: Change in Hemoglobin (HbA1c)
Description: HbA1c (percent) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens were analyzed at a central research laboratory
Time Frame: 12-month change from baseline fasting HbA1c
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: percentage of HbA1c in blood
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 66 | 55
percentage of HbA1c in blood | -0.2 [-0.2 to -0.1] | -0.1 [-0.1 to 0]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.083, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

11. Secondary Outcome: Change in Hemoglobin (HbA1c)
Description: HbA1c (percent) blood samples will be taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens are analyzed at central research laboratory
Time Frame: 24-month change from baseline fasting HbA1c
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: percentage of HbA1c in blood
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 56 | 44
percentage of HbA1c in blood | 0.0 [-0.1 to 0.1] | 0.1 [-0.0 to 0.1]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.778, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

12. Secondary Outcome: Change in Total Cholesterol
Description: Fasting total cholesterol (mg/dL) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens were analyzed at a central research laboratory.
Time Frame: 12-month change from baseline fasting total cholesterol
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 66 | 54
mg/dL | -6.2 [-11.6 to -0.8] | -6.1 [-13.9 to 1.7]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.982, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

13. Secondary Outcome: Change in Total Cholesterol
Description: as for outcome 12
Time Frame: 24-month change from baseline fasting total cholesterol
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 56 | 43
mg/dL | 4.1 [-3.1 to 11.4] | -7.2 [-18.6 to 4.2]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.081, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

14. Secondary Outcome: Change in High-density Lipoprotein (HDL)
Description: Fasting HDL (mg/dL) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens were analyzed at a central research laboratory.
Time Frame: 12-month change from baseline fasting HDL
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 54
mg/dL | 3.3 [1.2 to 5.4] | 2.8 [0.7 to 4.8]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.712, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

15. Secondary Outcome: Change in High-density Lipoprotein (HDL)
Description: as for outcome 14
Time Frame: 24-month change from baseline fasting HDL
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
Number analyzed (Participants) | 56 | 43
mg/dL | 3.5 [1.6 to 5.4] | 4.7 [2.7 to 6.8]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus 30-minute Calls vs Placebo Comparator: DPP Minimal 15-minute Calls; Test type: Superiority; p = 0.371, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

16. Secondary Outcome: Change in Low-density Lipoprotein (LDL)
Description: Fasting LDL (mg/dL) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens were analyzed at a central research laboratory.
Time Frame: 12-month change from baseline fasting LDL
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 53
mg/dL | -6.3 [-11.2 to -1.4] | -5.3 [-11.9 to 1.4]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.801, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

17. Secondary Outcome: Change in Low-density Lipoprotein (LDL)
Description: Fasting LDL (mg/dL) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens are analyzed at a central research laboratory.
Time Frame: 24-month change from baseline fasting LDL
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 56 | 43
mg/dL | 1.8 [-4.4 to 7.9] | -8.6 [-18.8 to 1.6]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.069, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

18. Secondary Outcome: Change in Triglycerides
Description: Fasting triglycerides (mg/dL) blood samples were taken by venipuncture after confirmed minimum overnight 8-hour fast. Specimens are analyzed at a central research laboratory.
Time Frame: 12-month change from baseline fasting triglycerides
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 53
mg/dL | -20.0 [-28.2 to -11.9] | -10.6 [-23.1 to 1.9]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.193, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

19. Secondary Outcome: Change in Triglycerides
Description: as for outcome 18
Time Frame: 24-month change from baseline fasting triglycerides at 24 months
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 56 | 43
mg/dL | -5.8 [-16.9 to 5.3] | -17.0 [-30.5 to -3.5]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.197, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

20. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: SBP (mmHg) measured by arm cuff digital blood pressure monitor (OMRON HEM90HXC)
Time Frame: 12-month change from baseline SBP
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 95 | 84
mmHg | -2.9 [-6.3 to 0.4] | -1.5 [-5.6 to 2.5]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.594, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

21. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: SBP (mmHg) measured by arm cuff digital blood pressure monitor (OMRON HEM90HXC)
Time Frame: 24-month change from baseline SBP
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 60
mmHg | 0.4 [-4.0 to 4.9] | -3.3 [-9.5 to 2.9]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.328, t-test, 2 sided

22. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: DBP blood pressure (mmHg) measured by arm cuff digital blood pressure monitor (OMRON HEM90HXC)
Time Frame: 12-month change from baseline DBP
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 95 | 84
mmHg | -4.5 [-6.3 to -2.7] | -3.3 [-5.6 to -0.9]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.398, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

23. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: DBP (mmHg) measured by arm cuff digital blood pressure monitor (OMRON HEM90HXC)
Time Frame: 24-month change from baseline DBP.
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 60
mmHg | -1.6 [-3.7 to 0.5] | -3.7 [-7.0 to -0.4]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.288, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

24. Secondary Outcome: Change in Physical Function
Description: Short Physical Performance Battery total score (0-12) includes three function tests (each scored 0-4) and summed.
  The subtests are (1) gait speed measured in meters/second on a 4-meter walk route; (2) 3 progressive standing balance tests; (3) 5 chair stands.
  Change in Total Score is reported here. Higher score indicates better physical function.
Time Frame: 12-month change from baseline on total score
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight with the exception of 1 participant in the Active Comparator and 2 participants in the Placebo Comparator who did not attempt the test due for physical safety reasons.
Measure: Mean (95% Confidence Interval); unit: units on a scale (higher is better)
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 94 | 82
units on a scale (higher is better) | 0.21 [-0.03 to 0.45] | 0.11 [-0.19 to 0.41]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.592, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

25. Secondary Outcome: Change in Physical Function
Description: as for outcome 24
Time Frame: 24-month change from baseline total score
Population: The analysis population corresponds to the that of the objectively measured primary outcome of bodyweight with the exception of 1 participant in the Placebo Comparator who did not attempt the test due for physical safety reasons.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 65 | 59
units on a scale | -0.12 [-0.53 to 0.29] | -0.05 [-0.44 to 0.33]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.805, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

26. Other Pre Specified Outcome: Change in Health Related Quality of Life
Description: Short-form 12-item health status questionnaire (SF-12) produces two scores; a physical component summary score (PCS) and a mental component summary score (MCS). Scores range from 0-100 with higher scores indicating better health related quality of life outcome. Each component score is transformed (standardized) using a mean of 50 and a standard deviation of 10. Scores below 50 suggest below average perceived health-related quality of life (e.g., a T-Score of 42 is indicative of a clinically relevant threshold for elevated depressive symptoms on the MCS scale).
Time Frame: 12-month change from baseline SF-12 score: PCS component and MCS component
Population: Note: We obtained mailed survey data from n = 1 additional subject in each of the Active Comparator and Placebo Comparator Groups who did not otherwise have an in-person clinic visit (for the weight primary outcomes) on which the Participant Flow diagram is based.
Measure: Mean (95% Confidence Interval); unit: T-scores
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 96 | 85
T-scores
  PCS Component Score | 1.0 [-0.7 to 2.6] | 1.9 [0.2 to 3.7]
  MCS Component Score | -0.1 [-1.7 to 1.6] | 0.5 [-1.3 to 2.4]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; The p value provided here is for the physical component summary score (PCS) only; Test type: Superiority; p = 0.421, t-test, 2 sided — The a priori threshold for significance is 0.05

27. Other Pre Specified Outcome: Change in Health Related Quality of Life
Description: Short-form 12-item health status questionnaire produces two scores; a physical component summary score (PCS) and a mental component summary score (MCS). Scores range from 0-100 with higher scores indicating better health related quality of life. Each component score is transformed (standardized) using a mean of 50 and a standard deviation of 10. Scores below 50 suggest below average perceived health-related quality of life (e.g., a T-Score of 42 is indicative of a clinically relevant threshold for elevated depressive symptoms on the MCS scale).
Time Frame: 24-month change from baseline SF-12 score: PCS and MCS
Population: Note: We obtained mailed survey data from n = 8 additional subjects in the Active Comparator Group, and n = 9 additional subjects in the Placebo Comparator Group who did not otherwise have an in-person clinic visit (for the weight primary outcomes) on which the Participant Flow diagram is based.
Measure: Mean (95% Confidence Interval); unit: T-scores
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 73 | 69
T-scores
  PCS Component | -0.4 [-2.2 to 1.3] | 1.5 [-0.6 to 3.7]
  MCS Component | -0.1 [-2.1 to 1.8] | -1.5 [-3.9 to 0.9]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority — The p value provided here is for the physical component summary score (PCS) only; p = 0.160, t-test, 2 sided

28. Other Pre Specified Outcome: Change in Mood
Description: The Center for Epidemiologic Studies Depression (CES-D) is a 20- item scale (scores range 0-60 with higher score indicating greater depressive symptoms). Scores should not be considered diagnostic, but they have been used to estimate the severity of depressive symptoms. Scores from 10-15 have been used to indicate mild depressive symptoms, 16-24 "moderate" or "significant" depressive symptoms, and >=25 "severe" depressive symptoms.
Time Frame: 12-month change from baseline CES-D
Population: Note: CES-D data was missing for n = 2 subjects in the Active Comparator Group (for whom we measured primary weight outcomes in person) and there was n = 2 additional subjects in the Placebo Comparator Group who had no in person weight measures but did submit CES-D data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 93 | 87
units on a scale | 0.8 [-0.6 to 2.2] | -0.5 [-1.8 to 0.9]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.196, t-test, 2 sided — The a priori threshold for significance is 0.05

29. Other Pre Specified Outcome: Change in Mood
Description: as for outcome 28
Time Frame: 24-month change from baseline CES-D
Population: Note: CES-D data was available for an additional n = 7 subjects in the Active Comparator Group and n = 11 additional subjects in the Placebo Comparator Group who otherwise had no in-person visit and primary outcome weight measures.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator: DPP Plus: 30-minute Calls | Placebo Comparator: DPP Minimal: 15-minute Calls
Number analyzed (Participants) | 72 | 71
units on a scale | -0.0 [-1.3 to 1.3] | 0.6 [-1.0 to 2.3]
Statistical Analysis 1: Comparison: Active Comparator: DPP Plus: 30-minute Calls vs Placebo Comparator: DPP Minimal: 15-minute Calls; Test type: Superiority; p = 0.532, t-test, 2 sided — The a priori threshold for statistical significance is 0.05

ADVERSE EVENTS:
Time Frame: Serious (SAE) and non-serious (AE) adverse event data were collected over the full study period of 24 months as reported to either independent assessment staff at the regular follow-up visits or ad-hoc to intervention staff at the time of phone conferences.
Description: We grouped adverse events by body or organ system, including "general disorders". Pregnancy, Puerperium and Perinatal Conditions were deemed N/A because of age. SAE and AE were collected and presented as follows: (1) The DPP Core Intervention (0-6 months) for ALL (N = 314) participants, and (2) The cumulative DPP Post-Core Intervention (7-24 months), categorized by two treatment arms DPP Plus: 30 Minute Calls (n =129) and DPP Minimal: 15 Minute Calls (n = 129).
Groups:
- Placebo Comparator: DPP Minimal 15-minute Calls: DPP Support 15-minute calls include no further behavioral intervention or self-monitoring material; phone contacts are unstructured and designed to promote peer support and accountability. Sessions occur once-per-month from months 7 to 12, and every-two-months from months 13 to 24.
Arm/Group | DPP Core Program | Active Comparator: DPP Plus 30-minute Calls | Placebo Comparator: DPP Minimal 15-minute Calls
All-Cause Mortality (participants affected / at risk) | 0/314 | 1/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 2/314 | 2/129 | 4/129
Other Adverse Events (participants affected / at risk) | 23/314 | 8/129 | 6/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DPP Core Program (N=314) | Active Comparator: DPP Plus 30-minute Calls (N=129) | Placebo Comparator: DPP Minimal 15-minute Calls (N=129)
Blood Cancer/Multiple Myeloma (Blood and lymphatic system disorders) | 0 | 1 | 0 — Plasma Cell Cancer, Multiple Myeloma
Subdural hematoma (Surgical and medical procedures) | 1 | 0 | 0 — Fell at home and hit head. Craniotomy performed.
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — In Situ Ductal Cell Breast Cancer
Covid-19 Hospitalization (Infections and infestations) | 0 | 0 | 1 — Extended Stay, Respirator Needed
Cancerous Neuroendocrine Tumor (Stomach) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — Endosopic Surgery to Remove 2 Tumors
Stroke (Vascular disorders) | 0 | 0 | 2 — Not otherwise specified
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Lung Cancer with Metastases to the Brain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DPP Core Program (N=314) | Active Comparator: DPP Plus 30-minute Calls (N=129) | Placebo Comparator: DPP Minimal 15-minute Calls (N=129)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 23 (23) | 8 (8) | 6 (6)

LIMITATIONS AND CAVEATS:
The study is likely underpowered for the primary outcome of weight change, due to recruitment targets not being met during the Covid-19 pandemic and greater than expected loss to follow-up for objective measurements in clinic (starting March 2020).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03500640/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03500640/SAP_001.pdf
  • Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT03500640/ICF_002.pdf